CLINICAL TRIAL: NCT04245358
Title: Open Non-Comparative Study To Evaluate The Performance And Safety Of The Medical Device Ainara® Vaginal Gel, In Post-Menopausal Women Affected By Vaginal Dryness
Brief Title: Open Non-Comparative Clinical Trial Study To Evaluate The Performance And Safety Of Ainara®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Italfarmaco (Industry)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMS/18/AINARA/02
Record Dates: First submitted 2020-01-27; First posted 2020-01-28 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2020-01

CONDITIONS: Vaginal Disease
MeSH Terms: conditions — Vaginal Diseases

STUDY DESIGN:
Intervention Model Description: Open-label, non-comparative, interventional multicenter study. The recently developed polycarbophilic, vaginal moisturizing gel (Ainara®) is widely used by gynaecologists in Europe to relieve vaginal dryness and related symptoms. Regarding the design choice, the adoption of a comparison versus placebo was not possible for technical reasons (the impossibility to use a real placebo without moisturizing effects).
  The Research Question of the present study is the following: in a population of post-menopausal women affected by vaginal dryness, will a 1-month treatment with polycarbophilic vaginal moisturizing gel (Ainara®) significantly decrease the symptomatology evaluated by VHI and VAS in comparison with the baseline condition?
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ainara (Other): Ainara is a class II medical device, already marketed in several EU countries. Each administration kit (subject kit) for patients of Ainara® will contain a box with 1 tube with 30 g gel, 1 cannula and 1 plunger. The gel quantity is enough for one subject over the course of the study (1 g at each administration).
  Interventions: Device: Ainara

INTERVENTIONS:
Device: Ainara — 1g of gel per administration

SUMMARY:
This study evaluates treatment with the medical device Ainara on the improvement of vaginal dryness evaluated by Vaginal Health Index (VHI) and Visual Analog Scale (VAS) in comparison with the baseline condition.

DETAILED DESCRIPTION:
Detailed Description: This is an open, non-comparative, multicenter study that evaluates the performance and safety of the medical device Ainara.

In this study the investigators use polycarbophilic vaginal moisturizing gel (Ainara) for symptomatic treatment of vaginal dryness and monitor its impact on vaginal dryness symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women (total cessation of menses for ≥ 1 year) according to the STRAW criteria, aged ≥ 50 to ≤ 70 years;
* Diagnosis of vaginal dryness by:

  * Subjective dryness, any objective sign of VVA, pH>5 as reported in the AGATA study
  * VHI < 15.
* Body mass index (BMI) ≥ 18.5 to ≤ 36 kg/m2;
* Able to communicate adequately with the Investigator and to comply with the requirements for the entire study.

Capable of and freely willing to provide written informed consent prior to participating in the study.

Exclusion Criteria:

* Malignancy (also leukemic infiltrates) within 5 years prior to Day 0 (except for treated basal cell/squamous cell carcinoma of the skin).
* Genital bleeding.
* Estrogen vaginal treatment during the study period (it was permitted only if terminated at least 6 months before study).
* Systemic estrogen therapy (it was permitted only if terminated at least 6 months before study).
* Subjects with illness, or other medical condition that, in the opinion of the investigator, would compromise participation or be likely to lead to hospitalization during the study or be likely to lead to hospitalization during the course of the study.
* Clinical evidence of acute infection currently requiring treatment (syphilis, herpes simplex, human papilloma virus, gonorrhea, chlamydia, lymphogranuloma venereum, etc.); clinical evidence or history of chronic infectious disease (i.e. tuberculosis).
* Psychosis, schizophrenia, mania, depressive disorders, history of suicide attempt or suicidal ideation, or any other psychiatric illness (except for intermittent anxiety).
* Known allergy to tested IMDs or its excipients.
* Drug or alcohol abuse in the 12 months prior to Day 0.
* Participation in an interventional clinical study or administration of any investigational agents in the previous 30 days.
* Presence of any clinically significant medical condition judged by the investigator to preclude the patient's inclusion in the study

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female have vagina so only female can have vagina disease.
Enrollment: 50 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Vaginal Health Index (VHI) | 30 days
  Vaginal Health Index: the changing from baseline to day 30 (final visit) for VHI mean value; The minim score is 5 and the maxim is is 25. For a patient to be included in study, the score must be lower than 15
Visual Analogue Scale (VAS) | 30 days
  Visual Analogue Scale: the changing from baseline to day 3, 7, 21, 30 (final visit) for VAS mean value; The minim score is 0 and the maxim score is 5, where 0 represents no symptoms and 3 represents severe symptoms

SECONDARY OUTCOMES:
subjective symptoms | 30 days
  • subjective symptoms: dryness, itching, burning, dyspareunia, and dysuria reported on patient diary and scored as reported in the AGATA study as follows: 0 = absence, 1 = slight, 2 = moderate, and 3 = severe intensity. The change in these variables will be evaluated from baseline to day 3, 7, 21, 30 (final visit).
objective signs in the vaginal mucosa | 30 days
  • objective signs in the vaginal mucosa: dryness, thinning rugae, pallor, fragility, and petechiae scored as reported in the AGATA study by Investigator as: 0 = absence, 1 = slight, 2 = moderate, and 3 = severe alteration. The change in these variables will be evaluated from baseline to 30 day (final visit).
Vaginal pH | 30 days
  • Vaginal pH: it will be measured by the Investigators with a test strip delivered by Sponsor. The baseline values can be ≥ 5.0 (this was the minimum value need for vaginal atrophy diagnosis in AGATA study) to 9.0. The Investigator will insert the pH strip into the upper wall of the vagina and will consider the reading made while the strip is still damp. The change in the mean value of this outcome will be evaluated from baseline to 30 day (final visit).
Vaginal Trophism Maturation Value (MV) | 30 days
  • Vaginal Trophism Maturation Value (MV): This outcome will be obtained from the cellular count of the vaginal smears at baseline and at the 30 days visit. The samples will be fixed, stored, and sent in the local laboratory in Timisoara, Romania (address details in TMF) for staining (Papanicolaou technique) and subsequent analysis. Samples will be evaluated by one independent cytopathologist blinded to the treatment. The MV will be calculated according to the following formula: MV = [1x (% superficial cells)] + [0.6x (% intermediate cells)] + [0.2x (% parabasal cells)]. The comparison will be between baseline and 30 days values.
Female Sexual Function Index (FSFI) | 30 days
  • Female Sexual Function Index (FSFI) Romanian version, evaluated by Investigator and analysed considering the change from baseline to 30 days (final visit).
Sexual Function (SF 12) | 30 days
  • SF 12 (Romanian version) evaluated by Investigator and analysed considering the changing from baseline to 30 day (final visit).
Global Symptom Score (GSS) | 30 days
  • Global Symptom Score (GSS) a composite score of symptoms, will be obtained to assess the effect of treatment on all individual symptoms taken as a whole. It will be calculated by the addition of the intensity scores of all individual symptoms (range, 1-15: 1 = only mild vaginal dryness, 15 = all five symptoms severe in intensity). This outcome will be compared, by assessing the change from baseline visit to 30 days visit (final visit).
Patient Global Assessment of Safety (PGAS) | 30 days
  • Patient Global Assessment of Safety (PGAS): it will be reported by the subject at all visits and all phone contacts in the patient diary using the 4-point scale:
  1= very good safety, 2 = good safety, 3 = moderate safety and 4 = poor safety.
Investigator Global Assessment of Safety (IGAS) | Time frame: 30 days
  • Investigator Global Assessment of Safety (IGAS): it will be reported by the Investigator using the 4-point scale:
  1= very good safety, 2 = good safety, 3 = moderate safety and 4 = poor safety. IGAS will be evaluated at the last visit, only.
AE, ADE, SAE, SADE | 30 days
  • AE, ADE, SAE, SADE: they will be reported by the Investigators according to the current legislation. All adverse events will be collected by Investigators at all visits and phone contacts and evaluated considering the change from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Liviu Cristian PĂTRAȘCU, MD, Principal Investigator — Fizio Center
Locations (1):
- Fizio Center, Timișoara, Timiș County, Romania

IPD SHARING:
Plan to Share IPD: No